CLINICAL TRIAL: NCT00871026
Title: Randomized Controlled Clinical Study Comparing Conventional and CAD/CAM-Based Treatment With Fixed Orthodontic Appliances
Brief Title: Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) - Based Planning and Creation of Orthodontic Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Paul-G. Jost-Brinkmann, Prof. Dr., Charité - Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JO 207/4-1-5
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Orthodontics
Keywords: CAD/CAM; orthodontics; fixed appliance; tooth movement; Adverse Effects; Time Factors; Treatment Outcome
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CAD/CAM group, customized archwires
  Interventions: Procedure: orthodontic treatment with customized archwires
- 2 (Active Comparator): prefabricated archwires (superelastic)
  Interventions: Procedure: orthodontic treatment with prefabricated archwires

INTERVENTIONS:
Procedure: orthodontic treatment with customized archwires — orthodontic treatment with customized archwires
  Other Names: SureSmile, CAD/CAM
  Arms: 1
Procedure: orthodontic treatment with prefabricated archwires — orthodontic treatment with prefabricated archwires
  Other Names: prefabricated archwires, conventional orthodontics
  Arms: 2

SUMMARY:
In orthodontics, conventional fixed appliances, usually consisting of prefabricated components, require step-by-step adjustment in order to move teeth in the planned direction.

May treatment be improved with customized archwires?

Study hypotheses:

* By using CAD/CAM in planning and fabrication of customized archwires, unnecessary tooth movements can be avoided and teeth can be moved on their direct path to the intended position.
* The application of CAD/CAM improves reproducibility, efficiency, and quality of orthodontic treatment.

DETAILED DESCRIPTION:
In orthodontics, conventional fixed appliances, usually consisting of prefabricated components, require step-by-step adjustment in order to move teeth in the planned direction. At the moment there is no tool, that allows to predict the treatment result. Using conventional orthodontic treatment methods the orthodontist approaches the final result using the trial-and-error-method, bending the wires in each appointment until both, patient and orthodontist are satisfied. Usually there is only a general treatment plan, but not a detailed treatment plan of each tooth movement. This leads to a longer treatment time and causes more costs. Besides the probability of side effects (such as caries root resorption) increases with the duration of the treatment.

In this case the chosen technology is called SureSmile(R)(by OraMetrix). SureSmile allows the collection 3D-data intraorally and from plaster models, it gives a possibility of computer aided treatment planing (Computer Aided Design) and the manufacturing of customized archwires (Computer Aided Manufacturing).

This new technology promises to reduce the time and effort of an orthodontic treatment providing predictability and quality also minimizing negative side effects.

This technology could - using this diagnostic 3D-system - help to understand orthodontic movement and basic principles of the remodeling of the periodontium and to improve orthodontic mechanics.

ELIGIBILITY:
Inclusion Criteria:

* treatment with fixed orthodontic appliances is indicated
* complete secondary dentition
* age: 11-30
* in good general health
* patient is informed about study and agrees to participate

Exclusion Criteria:

* syndromes affecting bones and teeth
* cleft lip and palate
* inflammation or reduction (more than 50%) of periodontium
* intake of drugs affecting tooth movement and bone formation
* disturbance of bone formation
* disturbance of thyroidal function
* pregnancy
* participation in additional study affecting oral hygiene
* former therapy with ionized radiation or cytostatic drugs
* caries (active phase)
* alcohol dependency

Ages: 11 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Duration of the orthodontic treatment (overall and every appointment) | every 6 weeks until the end of the treatment

SECONDARY OUTCOMES:
Quality measured using a quality index (ABO-Score)
Amount of root resorption comparing x-rays before and after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Georg Jost-Brinkmann, Prof, Study Chair — Charite - Universitätsmedizin
Locations (1):
- Department of Orthodontics, Dentofacial Orthopedics and Pedodontics, Charité - Universitätsmedizin Berlin, Berlin, Germany